CLINICAL TRIAL: NCT04157660
Title: Effect of Short-term Ambulatory Oxygen Therapy on Cardiopulmonary Exercise Capacity (CPET) in Patients With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Effect of Short-term Oxygen During CPET in HFpEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KEK-ZH-NR. 2012-0251_3
Record Dates: First submitted 2019-08-30; First posted 2019-11-08 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure, Diastolic (HFpEF)
MeSH Terms: conditions — Heart Failure; Heart Murmurs

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemental oxygen (Experimental): Supplemental oxygen will be applied via a mask during CPET
  Interventions: Procedure: Oxygen application
- Sham room air (Sham Comparator): Room air will be applied similarly to oxygen
  Interventions: Procedure: Sham room air

INTERVENTIONS:
Procedure: Oxygen application — Oxygen application Supplemental oxygen via mask
  Arms: Supplemental oxygen
Procedure: Sham room air — Room air will be applied via mask
  Arms: Sham room air

SUMMARY:
In a randomized, sham-controlled crossover trial the investigators will test whether supplemental oxygen given during cardiopulmonary exercise testing will improve exercise performance and physiological parameters in patients with heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF, stable medication for at least 4 weeks.

Exclusion Criteria:

* instable status, pregnancy, clinically relevant concomitant diseases, inability to follow the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Work Rate (Watt) | 1 day
  Maximal Work Rate (Watt max) measured during cardiopulmonary exercise test oxygen vs. room air
Endurance Time (s) | 1 day
  Endurance (s) with 75% Wmax measured during cardiopulmonary exercise test oxygen vs. room air

SECONDARY OUTCOMES:
Peak Oxygen uptake (VO2 max) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Respiratory Exchange Ratio (RER) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Changes in arterial blood parameters (pH) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Changes in arterial blood parameters (PaO2) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Changes in arterial blood parameters (PaCO2) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Changes in arterial blood parameters (Lactat) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Changes in arterial blood parameters (Bicarbonate) | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
muscle tissue oxygen | 1 day
  Oxygen Saturation in the muscle measured with near-infrared spectroscopy oxygen vs. room air
cerebral tissue oxygen | 1 day
  Oxygen Saturation in the brain measured with near-infrared spectroscopy oxygen vs. room air

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, Prof. Dr., Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muller J, Lichtblau M, Saxer S, Calendo LR, Carta AF, Schneider SR, Berlier C, Furian M, Bloch KE, Schwarz EI, Ulrich S. Effect of Breathing Oxygen-Enriched Air on Exercise Performance in Patients With Pulmonary Hypertension Due to Heart Failure With Preserved Ejection Fraction: A Randomized, Placebo-Controlled, Crossover Trial. Front Med (Lausanne). 2021 Jul 28;8:692029. doi: 10.3389/fmed.2021.692029. eCollection 2021. PMID 34395475